CLINICAL TRIAL: NCT00793312
Title: To Evaluate the 'Real World' Clinical Performance of the Medtronic Endeavor™ Zotarolimus Eluting Coronary Stent System in Chinese Patients, A Prospective, Multicenter Registry
Brief Title: China Endeavor Registry: A Registry With The Endeavor Zotarolimus Eluting Coronary Stent in China
Status: Completed | Type: Observational
Sponsor: Medtronic Vascular (Industry)
Collaborators: Medtronic Cardiovascular Asia Pacific (Industry)
Responsible Party: Sponsor
Other Study IDs: version 3.0 - 12 Nov 2008
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Last update posted 2012-10-17 (Estimated); Status verified 2012-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective is to document the acute and mid-term safety and overall clinical performance of the Endeavor(TM) Zotarolimus Eluting Coronary stent system in a "real world" Chinese patient population requiring stent implantation.

To assess the event rate in patient subgroups with specific clinical indications and/or vessel or lesion characteristics.

DETAILED DESCRIPTION:
The safety and efficacy of the Endeavor(TM) Zotarolimus Eluting Coronary Stent System has been assessed in a series of studies, e.g. ENDEAVOR I and ENDEAVOR II. The stent is composed of a cobalt alloy and is coated with a proprietary drug compound zotarolimus that is designed to reduce restenosis.

This registry with the Endeavor(TM) Zotarolimus Eluting Coronary Stent System is being initiated 1) to expand the clinical knowledge base by including 'real world'patients in China and 2) to assess the event rate in Chinese patients known to have a higher risk of major adverse cardiac events, for example patients with diabetes mellitus, small vessels and long lesions.

In total the plan is to enroll about 2200 patients from 37 sites.

Follow-up will be one year for the main patients with cohort to collect acute and mid-term follow-up data, but will be extended to two years for certain patient subgroups.

ELIGIBILITY:
Inclusion Criteria:

* Patient is > 18 years of age (or minimum age as required by local regulations).
* The patient has consented to participate by signing the "Patient Informed Consent Form" and/or has authorized the collection and release of his medical information by signing the "Patient Data Release Consent Form".
* Patient is suitable for implantation of one or more Endeavor™ Zotaroliums Eluting Coronary Stent System in one or more native artery target lesions.
* Patient indication, lesion length and vessel diameter of the target lesion(s) are according to the Indications for Use' as mentioned in the 'Instructions for Use' that comes with every Endeavor™ Zotarolimus Eluting Coronary Stent System.
* The patient is willing and able to cooperate with registry procedures and required follow up

Exclusion Criteria:

* Women with known pregnancy or who are lactating.
* Patients with hypersensitivity or allergies to aspirin, heparin, clopidogrel, ticlopidine, drugs such as zotaroliums, rapamycin, tacrolimus, sirolimus or similar drugs, or any other analogue or derivative, cobalt, chromium, nickel, molybdenum or contrast media.
* Patients in whom anti-platelet and/or anticoagulation therapy is contraindicated.
* Patients who are judged to have a lesion that prevents complete inflation of an angioplasty balloon.
* Current medical condition with a life expectancy of less than 12 months.
* The subject is participating in another device or drug study. Subject must have completed the follow-up phase of any previous study at least 30 days prior to enrollment in this trial. The subject may only be enrolled in this Registry once.
* Patients with medical conditions that preclude the follow-up as defined in the protocol or that otherwise limits participation in this registry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an indication for coronary stent implantation according to the 'Instructions for Use' of the Endeavor™ Zotarolimus Eluting Coronary Stent System, or at investigators' discretion. All consecutive patients who receive one or more Endeavor™ stents in one or more target lesions should be included.
Sampling Method: Probability Sample
Enrollment: 2210 (Actual)
Dates: Start 2007-11; Primary Completion 2009-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
MACE | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Jiyan Chen, Professor, Principal Investigator — Guangdong Provincial People's Hospital; Yaling Han, Professor, Principal Investigator — Shenyang North Hospital; Yong Huo, Professor, Principal Investigator — Peking University First Hospital; Weimin Wang, Professor, Principal Investigator — Beijing People's Hospital; Bo Xu, Director, Principal Investigator — Fu Wai Hospital, Beijing, China